CLINICAL TRIAL: NCT07273929
Title: Multicenter Randomised Controlled Trial: Benefit of Intra-pocket Echo-guided Axillary Puncture Compared With Percutaneous Echo-guided Axillary Puncture and Cephalic Vein Dissection for the Primary Implantation of Intracardiac Electronic Devices.
Brief Title: Comparative Study of the Effectiveness of Three Access Routes for Implanting an Electronic Intracardiac Device
Acronym: MultiPM-ACCESS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL24_0743
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Primary Implantation of an Intracardiac Electronic Device Indication
Keywords: venous access; intracardiac device; ryhthmology

STUDY DESIGN:
Intervention Model Description: Multicenter randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 : Cephalic vein dissection (Experimental): After an incision in the deltopectoral groove and careful dissection of the superficial fatty layer, the cephalic vein is revealed and separated from its tissue attachments over a distance of approximately 2 centimetres before being cannulated in order to introduce the necessary guides.
  The electronic device will be fitted using the guides introduced in this way.
  Interventions: Procedure: Intervention 1: Cephalic vein dissection
- Group 2 : Percutaneous echo-guided axillary route (Experimental): A standard vascular linear ultrasound probe is placed in a single-use sterile sheath. The probe is brought into contact with the skin and the investigators then perform a needle puncture of the vein under ultrasound control. Once the puncture or punctures have been successful, a guide is inserted into the vein and the incision is made after the puncture.
  The electronic device will be fitted using the guides introduced in this way.
  Interventions: Procedure: Intervention 2 : Percutaneous echo-guided axillary route
- Group 3 : Intrapocket ultrasound-guided axillary route (Experimental): A special ultrasound probe (shaped like a hiccup) is placed in a single-use sterile sheath. After making an incision in the deltopectoral groove and dissecting the fatty layer, the probe is placed in contact with the pectoral muscle to visualise the axillary vein. Needle puncture of the vein is performed under ultrasound guidance. Once the puncture is successful, a guide is inserted into the vein.
  Interventions: Procedure: Intervention 3 : Intrapocket ultrasound-guided axillary route

INTERVENTIONS:
Procedure: Intervention 1: Cephalic vein dissection — After an incision in the deltopectoral groove and careful dissection of the superficial fatty layer, the cephalic vein is revealed and separated from its tissue attachments over a distance of approximately 2 centimetres before being cannulated in order to introduce the necessary guides.
  The electronic device will be fitted using the guides introduced in this way.
  Arms: Group 1 : Cephalic vein dissection
Procedure: Intervention 2 : Percutaneous echo-guided axillary route — A standard vascular linear ultrasound probe is placed in a single-use sterile sheath. The probe is brought into contact with the skin and we then perform a needle puncture of the vein under ultrasound control. Once the puncture or punctures have been successful, a guide is inserted into the vein and the incision is made after the puncture.
  The electronic device will be fitted using the guides introduced in this way.
  Arms: Group 2 : Percutaneous echo-guided axillary route
Procedure: Intervention 3 : Intrapocket ultrasound-guided axillary route — A special ultrasound probe (shaped like a hiccup) is placed in a single-use sterile sheath. After making an incision in the deltopectoral groove and dissecting the fatty layer, the probe is placed in contact with the pectoral muscle to visualise the axillary vein. Needle puncture of the vein is performed under ultrasound guidance. Once the puncture is successful, a guide is inserted into the vein.
  The electronic device will be fitted using the guides introduced in this way.
  Arms: Group 3 : Intrapocket ultrasound-guided axillary route

SUMMARY:
The implantation of an intra-cardiac electronic device (ICD) (pacemaker or defibrillator) is a frequent procedure, and one whose incidence is on the rise in the field of cardiology. In France in 2016, 69042 pacemakers and 8174 defibrillators were implanted.

The procedure involves inserting one or more intra-cardiac leads using venous access. Navigation in the heart chambers is guided by fluoroscopy. Each lead is connected to a box that is placed under the skin in the deltopectoral groove.

The venous vascular approach or venous access is a key stage. It can be time-consuming and a source of complications (haematoma, pneumothorax, nerve damage, catheter malfunction).

There are several methods of vascular access: cephalic vein dissection, subclavian vein puncture guided by anatomical landmarks, axillary puncture guided by scopy (X-rays) or intraoperative ultrasound.

The implantation of an intra-cardiac electronic device (ICD) (pacemaker or defibrillator) is a frequent procedure, and one whose incidence is on the rise in the field of cardiology. In France in 2016, 69042 pacemakers and 8174 defibrillators were implanted.

The procedure involves inserting one or more intra-cardiac leads using venous access. Navigation in the heart chambers is guided by fluoroscopy. Each lead is connected to a box that is placed under the skin in the deltopectoral groove.

The venous vascular approach or venous access is a key stage. It can be time-consuming and a source of complications (haematoma, pneumothorax, nerve damage, catheter malfunction).

There are several methods of vascular access: cephalic vein dissection, subclavian vein puncture guided by anatomical landmarks, axillary puncture guided by scopy (X-rays) or intraoperative ultrasound.

The most commonly used venous access for DEIC implantation in Europe today is cephalic vein dissection (60%). The subclavian vein is used in 21% of cases and the axillary vein in 19%.

There is currently no recommendation as to which technique should be used as first-line treatment.

The subclavian route is performed by puncture without direct visualisation of the vein, and therefore presents a risk of complications such as pneumothorax.

The cephalic route has few complications, but requires lengthy and tedious dissection and considerable experience. According to the literature, the failure rate is between 20 and 30%.

For axillary vein puncture, several options have been described: blind, scopy-guided with venography and ultrasound-guided.

Ultrasound-guided axillary puncture has been proposed for several years, but is currently not widely used. According to the literature, this technique seems to have a high success rate with a low complication rate, particularly with regard to the risk of pneumothorax. There are currently two ultrasound-guided axillary puncture techniques.

The 'intra-pocket' axillary puncture technique involves performing a puncture after making the incision using a special ultrasound probe (shaped like a golf club), placed in contact with the pectoral muscle.

Percutaneous" axillary puncture, on the other hand, is performed using a standard linear vascular ultrasound probe. Here the puncture is performed before the incision and the probe is placed in contact with the skin.

According to the literature currently available, the ultrasound-guided 'intra-pocket' technique appears to have a better success rate than the ultrasound-guided 'percutaneous' technique (95-99% success rate vs. 90-95%).

The investigators recently conducted the ACCESS study, a prospective, single-centre, randomised, open-label study comparing echo-guided 'intra-pocket' axillary puncture with the conventional cephalic vein dissection technique. the investigators demonstrated that this technique has a higher success rate than cephalic vein dissection, with a significant time saving (success rate: 99 vs. 87% (p=0.01), procedure time: 33.8 vs. 46.9 min,p= 0.005).

Our project is therefore to carry out a multicentre randomised trial to confirm these promising initial results and to assess the efficacy and safety of 'intra-pocket' echo-guided axillary venipuncture compared with 'percutaneous' echo-guided axillary venipuncture and the reference technique of cephalic dissection during implantation of a DEIC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* First implantation of a pacemaker or defibrillator (single or double chamber) or implantation of a lead in the left branch area in the case of a venticular lead.
* Informed consent signed by the patient

Exclusion Criteria:

* Implantation of an intra-cardiac triple-chamber electronic device (cardiac resynchronisation)
* Prior impossibility of venous access
* Pregnant, parturient or breast-feeding women
* Persons deprived of their liberty by judicial or administrative decision
* Persons under psychiatric care
* Persons admitted to a health or social establishment for purposes other than research
* Adults under legal protection (guardianship, curatorship)
* Persons not affiliated to a social security scheme or beneficiaries of a similar scheme
* Patients participating in other research that may interfere with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Success rates of the three procedures | During the intervention
  To assess the efficacy of echo-guided axillary puncture using the intra-pocket technique compared with the other 2 techniques in adult patients undergoing primary implantation of an intra-cardiac electronic device.
  The three groups were compared on the binary criterion of failure/success of access directly during the procedure. The success of the vascular approach is defined by the success rate of insertion of all the leads using the first venous access technique assigned by randomisation.

SECONDARY OUTCOMES:
Vascular access time | During the intervention
  Comparison between groups of vascular access time (superior vena cava time) measured in seconds: Time between skin incision and presence of all necessary guides in the superior vena cava for the 'intra pocket' axillary group and cephalic vein dissection / Time between first puncture and presence of all necessary guides in the superior vena cava for the 'percutaneous' axillary group.

OTHER OUTCOMES:
Total procedure time | During the intervention
  Comparison between groups of total procedure time measured in seconds: Time from skin incision to complete closure of scar for the 'intra-pocket' axillary puncture and cephalic vein dissection group / Time from first puncture to skin closure for the 'percutaneous' axillary group.
Exposure to ionising radiation time | During the intervention
  Comparison between groups of duration of exposure to ionising radiation measured in seconds.
Intensity of exposure to ionising radiation | During the intervention
  Comparison between groups of intensity of exposure to ionising radiation measured in mGray/cm2, during the procedure.
Intra-operative, post-operative and 3-month complications | Between inclusion and 3 months follow-up
  Comparison between groups of intra-operative complications, post-operative complications at 3 months of the operation including:
  * Nerve damage
  * Major loge haematoma (need for evacuation, transfusion required, prolongation of hospital stay)
  * Pneumothorax
  * Haemothorax
  * Pericardial effusion
  * Catheter displacement (requiring re-operation for replacement) Venous thrombosis
Occurrence of device infection (device infection or infective endocarditis requiring removal of the device) | Between inclusion and 3 months follow-up
  Occurrence of device infection (device infection or infective endocarditis requiring removal of the device)

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hôpital F. MITTERRAND, Dijon
  - Lyon-Croix Rousse, Lyon
  - Lyon-Louis Pradel, Lyon
  - Hôpital privé Jacques Cartier, Massy
  - CH Annexy-Genevois, site Annecy, Metz
  - CHU de Saint Etienne - Hôpital Nord, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No